CLINICAL TRIAL: NCT04480619
Title: Safety and Efficacy of Ga-68-IAC Positron Emission Tomography (PET/CT) for Diagnosis and Clinical Management in Metastatic Breast Cancer Patients.
Brief Title: Safety and Efficacy of Ga68-IAC PET/CT for Diagnosis and Clinical Management in Metastatic Breast Cancer Patients
Acronym: Shiva
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Advanced Imaging Projects, LLC (Industry)
Collaborators: All India Institute of Medical Sciences (Other); Post Graduate Institute of Medical Education and Research, Chandigarh (Other); University of Witwatersrand, South Africa (Other); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 145314
Record Dates: First submitted 2020-06-30; First posted 2020-07-21 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Angiogenic Breast Cancer

STUDY DESIGN:
Intervention Model Description: Ga-68-AC PET/CT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ga-68-IAC PET/CT (Experimental): Companion Ga-68 PET diagnostic for tumor targeted therapy
  Interventions: Diagnostic Test: Ga-68-IAC

INTERVENTIONS:
Diagnostic Test: Ga-68-IAC — Clinical management and diagnosis of Metastatic Breast Cancer.
  Other Names: Ga-68-IAC PET/CT

SUMMARY:
This is a phase I/IIa, open label, multicenter interventional study of Gallium-68 radiolabeled Integrin Adhesion Complex antagonist conjugate (Ga-68-IAC) Positron Emission Tomography (PET/CT) imaging, intended for diagnosis, and clinical management of patients with Metastatic breast cancer.

DETAILED DESCRIPTION:
This is a prospective non blinded trial, Phase I/IIa, multicenter, study in a total of up to 25 subjects with angiogenic therapy indication for breast cancer. All patients with confirmed diagnoses will undergo [18F]Fluoro-deoxyglucose (18F-FDG) PET/CT (6-12 mCi) and Ga-68-IAC PET/CT 2-5 mCi to evaluate safety, biodistribution, and response to treatment in metastatic breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with solid tumors (either 3+ by immunohistochemistry or with evidence of gene amplification (>2.0) by fluorescence in situ hybridization (FISH))

  * At least 18 years of age
  * Able to provide informed consent.

Karnofsky score greater than 50

* Females of childbearing potential must have a negative pregnancy test at screening/baseline
* AIP-301 Ga-68 positive scan define by SUV greater than 10.
* Adequate organ function, defined as:

  1. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L.
  2. Hemoglobin (Hb) ≥9 g/dl (transfusion or use of EPO is permitted).
  3. Platelets > 100,000/mm3
  4. Creatinine ≤ 1.5 x normal value based on the Cock Gault (CG) equation.
  5. AST or ALT ≤ 2.5 x ULN (or ≤5 x ULN in case of liver metastasis)
  6. Alkaline phosphatase ≤2.5 x ULN. Alkaline phosphatase may be more than 2.5 x ULN only in the case of bone metastases, and AST and ALT less than 1.5 x ULN.
  7. Total bilirubin ≤1.5 mg/dl (higher bilirubin levels are permitted if the patient has Gilbert's syndrome).

Baseline LVEF ≥50% measured using echocardiogram or equilibrium

isotopic ventriculography (MUGA).

Exclusion Criteria:

* • Serum creatinine >3.0 mg/dL (270 μM/L)

  * Hepatic enzyme levels more than 5 times upper limit of normal.
  * Known severe allergy or hypersensitivity to IV radiographic contrast.
  * Use of any other investigational product or device within 30 days prior to dosing or known requirement for any other investigational agent prior to completion of all scheduled study assessments.
  * Patients with a body weight of 400 pounds or more or not able to enter the bore of the PET/CT scanner due to BMI, because of the compromise in image quality with CT, PET/CT and MRI that will result.
  * Inability to lie still for the entire imaging time (e.g. cough, severe arthritis, etc.).
  * Inability to complete the needed investigational and standard-of-care imaging examinations due to other reasons (severe claustrophobia, radiation phobia, etc.)
  * Recognized concurrent active infection (e.g., HIV)
  * Previous Grade 3 or higher allergic reaction to Trastuzumab that resulted in discontinuation of Trastuzumab therapy. Any additional medical condition, serious intercurrent illness, or other extenuating circumstance that, in the opinion of the Investigator, may significantly interfere with study compliance.

    * Adult patients who require monitored anesthesia for PET scanning

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-10-30 (Estimated); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Specific Aims 1:To evaluate the safety, toxicity profile and tolerability of Ga-68-IAC in patients diagnosed with angiogenic breast cancer. | 6 Months
  Assess drug safety and tolerability measuring Incidence of adverse events. NCI Common Terminology Criteria for Adverse Events v5.0, where: Grade 1, mild; Grade 2, moderate; Grade 3, severe; Grade 4, life-threatening
Specific Aims 2:To evaluate biodistribution and dosimetry of Ga-68-IAC | 6 Months
  Assess drug safety and tolerability measuring incidence of abnormal vital signs. Vital signs will include measurements of respiratory rate, pulse rate, and systolic and diastolic blood pressure.
Specific Aims 3: To determine the recommended phase 2 dose (RP2D) of Ga-68-IAC examination | 6 Months
  Assess drug safety and tolerability measuring incidence of abnormal physical examination findings. Physical examination will be summarized for each body system such as head, eyes, ears, nose, and throat, and cardiovascular, dermatological, musculoskeletal, respiratory, gastrointestinal, genitourinary, and neurological systems.

SECONDARY OUTCOMES:
Specific Aim 1: To determine the pharmacokinetic and pharmacodynamic profile of Ga-68-IAC | 6 Months
  Assess drug uptake using median and maximum standardized uptake values (SUV).

CONTACTS AND LOCATIONS:
Locations (3):
- India (2):
  - Postgraduate Institute of Medical and Research, Chandigarh
  - All India Institute of Medical Sciences, New Delhi
- University of Witwatersrand, Johannesburg, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Data will be available after completion of clinical trial
Supporting Information: CSR
Time Frame: 2 years

REFERENCES:
- [Result] Baum RP, Kulkarni HR, Muller D, Satz S, Danthi N, Kim YS, Brechbiel MW. First-In-Human Study Demonstrating Tumor-Angiogenesis by PET/CT Imaging with (68)Ga-NODAGA-THERANOST, a High-Affinity Peptidomimetic for alphavbeta3 Integrin Receptor Targeting. Cancer Biother Radiopharm. 2015 May;30(4):152-9. doi: 10.1089/cbr.2014.1747. PMID 25945808
- [Result] Kim YS, Nwe K, Milenic DE, Brechbiel MW, Satz S, Baidoo KE. Synthesis and characterization of alphavbeta(3)-targeting peptidomimetic chelate conjugates for PET and SPECT imaging. Bioorg Med Chem Lett. 2012 Sep 1;22(17):5517-22. doi: 10.1016/j.bmcl.2012.07.024. Epub 2012 Jul 14. PMID 22853992